CLINICAL TRIAL: NCT04311684
Title: Development and Validation of Hybrid Brillouin-Raman Spectroscopy for Non-invasive Assessment of Mechano-chemical Properties of Urine Proteins as Biomarkers of Kidney Diseases
Brief Title: Non-invasive Assessment of Mechano-chemical Properties of Urine Proteins by Hybrid Brillouin-Raman Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nazarbayev University (Other)
Collaborators: National Scientific Medical Center, Kazakhstan (Other Government); Astana Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 091019CRP2105
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Nephrotic Syndrome
Keywords: urinary proteins; Brillouin spectroscopy; surface enhanced Raman spectroscopy; proteomics; non-invasive assessment
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with proteinuria: Patients with newly diagnosed glomerulonephritis with different range of proteinuria at the age between 18-65 years and estimated glomerular filtration rate (GFR) ≥60 ml/min will be included for urine protein measurements
  Interventions: Device: hybrid Brillouin-Raman spectroscopy
- Healthy volunteers: Healthy men/women between age group 18-65 years will be included for urine protein measurements
  Interventions: Device: hybrid Brillouin-Raman spectroscopy

INTERVENTIONS:
Device: hybrid Brillouin-Raman spectroscopy — Combination of Brillouin and surface-enhanced Raman (SERS) spectroscopy for assessment of both visco-elastic (i.e. mechanical) and chemical characterization of urinary proteins at the same time from the same excitation laser source

SUMMARY:
The proteinuria is widely recognized as a marker of kidney disease severity, as well as the predictor of renal function decline, cardiovascular outcomes, and all-cause mortality. However, the severity of kidney disease progression and these outcomes differs among patients with various amount of proteinuria. The potential mechanism underlining this disparity may be relevant to the quality and quantity of filtered proteins, especially their mechano-chemical properties such as physical viscosity and stiffness, amino-acid sequence, and molecular weight (low, middle and high molecular weight proteins). The goal of the current project is to develop and validate combined Brillouin & Surface-Enhanced Raman Scattering (SERS) Spectroscopy technique for simultaneous non-contact assessment of visco-elastic and chemical properties of urine proteins as biomarkers of kidney disease. Systematic studies of these properties of proteins in urine samples to be taken from diseased and healthy subjects will be cross-validated by Liquid Chromatography-Mass Spectrometry (LCMS). The project ultimately aims for the development of an optical spectroscopic sensor for rapid, non-contact monitoring of urine samples from patients in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients with any ethnic group, aged between 18-65 years old
* Newly diagnosed patients with glomerulonephritis and different range of proteinuria

Exclusion Criteria:

* patients aged <18 and >65 years,
* eGFR<60 ml/min,
* pregnant females,
* patients with diabetes mellitus, cancer, infectious diseases, and other life-treating comorbidities/conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The proposed study will include 20 healthy subjects and age/gender matched 80 patients with newly diagnosed glomerulonephritis with different range of proteinuria at the age between 18-65 years and estimated glomerular filtration rate (GFR) ≥60 ml/min. Exclusion criteria will be patients aged <18 and >65 years, eGFR<60 ml/min, pregnant females, patients with diabetes mellitus, cancer, infectious diseases and other life-treating comorbidities/conditions.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Non-invasive assessment of mechano-chemical properties of urine proteins by hybrid Brillouin-Raman spectroscopy in a patient with nephrotic syndrome | four weeks
  Urine sample measurements by Brillouin and surface enhanced Raman (SERS) spectroscopy

SECONDARY OUTCOMES:
Non-invasive assessment of mechano-chemical properties of urine proteins by hybrid Brillouin-Raman spectroscopy in a patient with nephrotic syndrome | four weeks
  Correlation and cross-validation of urinary protein Brillouin and SERS spectroscopy measurements by Liquid Chromatography-Mass Spectrometry (with proteomic measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Abduzhappar Gaipov, MD, PhD, Principal Investigator — Nazarbayev University School of Medicine
Locations (1):
- Nazarbayev University School of Medicine, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ikramova SB, Utegulov ZN, Dikhanbayev KK, Gaipov AE, Nemkayeva RR, Yakunin VG, Savinov VP, Timoshenko VY. Surface-Enhanced Raman Scattering from Dye Molecules in Silicon Nanowire Structures Decorated by Gold Nanoparticles. Int J Mol Sci. 2022 Feb 26;23(5):2590. doi: 10.3390/ijms23052590. PMID 35269733
- [Result] Aitekenov S, Sultangaziyev A, Abdirova P, Yussupova L, Gaipov A, Utegulov Z, Bukasov R. Raman, Infrared and Brillouin Spectroscopies of Biofluids for Medical Diagnostics and for Detection of Biomarkers. Crit Rev Anal Chem. 2023;53(7):1561-1590. doi: 10.1080/10408347.2022.2036941. Epub 2022 Feb 14. PMID 35157535
- [Result] Aitekenov S, Gaipov A, Bukasov R. Review: Detection and quantification of proteins in human urine. Talanta. 2021 Feb 1;223(Pt 1):121718. doi: 10.1016/j.talanta.2020.121718. Epub 2020 Oct 14. PMID 33303164
- [Result] Gaipov A, Utegulov Z, Bukasov R, Turebekov D, Tarlykov P, Markhametova Z, Nurekeyev Z, Kunushpayeva Z, Sultangaziyev A. Development and validation of hybrid Brillouin-Raman spectroscopy for non-contact assessment of mechano-chemical properties of urine proteins as biomarkers of kidney diseases. BMC Nephrol. 2020 Jun 15;21(1):229. doi: 10.1186/s12882-020-01890-x. PMID 32539773
- [Result] Gaipov A, Makhammajanov Z, Dauyey Z, Markhametova Z, Mussina K, Nogaibayeva A, Kozina L, Auganova D, Tarlykov P, Bukasov R, Utegulov Z, Turebekov D, Soler MJ, Ortiz A, Kanbay M. Urinary Protein Profiling for Potential Biomarkers of Chronic Kidney Disease: A Pilot Study. Diagnostics (Basel). 2022 Oct 25;12(11):2583. doi: 10.3390/diagnostics12112583. PMID 36359427
- See also: Project Details — https://research.nu.edu.kz/en/projects/development-and-validation-of-hybrid-brillouin-raman-spectroscopy